CLINICAL TRIAL: NCT03888378
Title: A Multi-Center, Double-Masked, Randomized, Vehicle-Controlled Study of the Efficacy and Safety of HY02 Ointment in Subjects With Inflamed Meibomian Gland Dysfunction
Brief Title: Study to Evaluate the Safety and Efficacy of Minocycline Ointment in Subjects With Inflamed Meibomian Gland Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hovione Scientia Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HY02-002
Record Dates: First submitted 2019-03-22; First posted 2019-03-25 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Meibomian Gland Dysfunction; MGD-Meibomian Gland Dysfunction
Keywords: Minocycline Topical; Tetracycline; Doxycycline; MGD; Meibomian Gland Disorder; Anti-Bacterial Agent; Anti-imflammatory Agent; Minocycline
MeSH Terms: conditions — Meibomian Gland Dysfunction; cyclopia sequence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Care provider is a designated dosing coordinator who will be unblinded for this study. Both participant and investigator will be blinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 0.3% Topical Minocycline Ointment (Active Comparator): Topical administration of 0.3% Topical Minocycline Ointment. Regimen: Apply BID (twice daily), morning and evening to eyelid margin
  Interventions: Drug: 0.3% Topical Minocycline Ointment
- 1% Topical Minocycline Ointment (Active Comparator): Topical administration of 1% Topical Minocycline Ointment. Regimen: Apply BID (twice daily), morning and evening to eyelid margin
  Interventions: Drug: 1% Topical Minocycline Ointment
- Topical Vehicle Ointment (Placebo Comparator): Topical administration of Topical Vehicle Ointment. Regimen: Apply BID (twice daily), morning and evening to eyelid margin
  Interventions: Other: Topical Vehicle Ointment

INTERVENTIONS:
Drug: 0.3% Topical Minocycline Ointment — 0.3% Topical Minocycline ointment to treat inflamed Meibomian Gland Dysfunction
  Other Names: HY02 Topical Ointment, 0.3%
  Arms: 0.3% Topical Minocycline Ointment
Drug: 1% Topical Minocycline Ointment — 1% Topical Minocycline ointment to treat inflamed Meibomian Gland Dysfunction
  Other Names: HY02 Topical Ointment, 1%
  Arms: 1% Topical Minocycline Ointment
Other: Topical Vehicle Ointment — Topical vehicle ointment to treat inflamed Meibomian Gland Dysfunction
  Other Names: HY02 Topical Ointment, 0%
  Arms: Topical Vehicle Ointment

SUMMARY:
To evaluate the efficacy and safety of two strengths of HY02 Ointment versus Vehicle administered twice daily for twelve weeks in subjects with a diagnosis of Inflamed Meibomian Gland Dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* At Visit 1, individuals of any gender or any race will be eligible for study participation if they:

  1. Have provided written informed consent prior to any study procedures.
  2. Are 18 years of age or above.
  3. Have a clinical diagnosis of moderate to severe MGD and who meet the following criteria, in a qualifying eyelid, at both Visit 1 (Screening) and Visit 2 (Randomization) examinations:

     1. Clinical sign severity score of at least 2 (moderate) on vascular engorgement at the eyelid margin and
     2. Clinical sign severity score of at least 2 (moderate) on plugging of the meibomian glands.
     3. Eye Discomfort Symptom score of ≥ 40 using VAS (0-100 point scale)
  4. Meet the following criteria, in a qualifying eye (same eye that qualifies for Inclusion #3), at both the Visit 1 (Screening) and Visit 2 (Randomization) examinations:

     1. Fluorescein corneal staining (FCS) total score ≥ 3 in the inferior, central, and nasal region combined score (NEI/Industry Workshop sections 1, 4 and 5 with 0-9 scale)
     2. Schirmer score of >7 mm without topical anesthesia
  5. Are willing and able to follow instructions and can be present for the required study visits for the duration of the study.
  6. Have a BCVA, using corrective lenses if necessary, in both eyes of at least +0.7 as assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) or modified ETDRS.
  7. If female, are non-pregnant, non-lactating and women of childbearing potential (WOCBP) must be using an acceptable method of birth control [e.g., an Intrauterine Contraceptive Device (IUCD) with a failure rate of <1%, hormonal contraceptives, or a barrier method] for the duration of the study. If a female subject is currently abstinent, they must agree to use one of the acceptable methods of birth control before they become sexually active.

Exclusion Criteria:

In order for subjects to be eligible at Visit 1 they may not:

1. Have presence of inflammation and/or active structural change in the iris or anterior chamber.
2. Have lid structural abnormalities such as entropion or ectropion.
3. In the eyelid that qualifies (based on Inclusion #3), have grade level 4 (Obstructed) on Character of Secretion of Meibomian Glands or grade level 4 (No glands are expressible) on the Expressibility of Meibomian Glands.
4. Subjects with ocular inflammatory conditions (e.g., conjunctivitis, keratitis, anterior blepharitis, etc.) not related to MGD.
5. Subjects who have FCS total score = 15 or a score = 3, in either eye, in the superior region NEI/Industry Workshop scale or subjects who have FCS with diffuse confluent staining, filaments or frank epithelial defects.
6. Have suspected ocular fungal, viral or bacterial infection.
7. Have had penetrating intraocular surgery in the past 90 days or require penetrating intraocular surgery during the study.
8. Have had ocular surface surgery within 12 months of Visit 1 (e.g., LASIK, refractive, pterygium removal).
9. Subjects who within the past 90 days have had cauterization of the punctum or changes to the status (insertion or removal) of punctal plug(s) before the Screening Visit.
10. Have used topical ocular or oral antibiotics within 30 days of the study or expect to use during the study.
11. Have used LipiFlow or hypochlorous acid spray within 30 days of the study or expect to use during the study.
12. If using inhaled or intranasal corticosteroids, unable to maintain a stable dose for the duration of the study.
13. Have ever used isotretinoin.
14. If using Omega-3 supplements, dose must be stable for 3 months prior to Visit 1 and for the duration of the study.
15. Have used topical cyclosporine within 30 days of the study or during the study.
16. Have used topical lifitegrast within 30 days of the study or during the study.
17. Have used systemic corticosteroids within 30 days prior to study entry or during study participation.
18. Have used topical ocular corticosteroids or ocular non-steroidal anti-inflammatory drugs (NSAIDs) within 30 days prior to study entry and during study participation.
19. Have used topical ocular antihistamine and/or mast cell stabilizers within 30 days prior to study entry or during study participation.
20. Are unable or unwilling to discontinue using any preserved or unpreserved topical ocular medications (including artificial tears) upon Screening and for the duration of the study.
21. Are unwilling to discontinue use of contact lenses during the study.
22. Are unwilling to discontinue use of cosmetic makeup applied to the eyelids or eye lashes at the Screening Visit and during the study. If makeup was used, it should be removed at least 12 hours prior to Visit 1.
23. Have a known hypersensitivity to minocycline, any other tetracycline antibiotic, or to any of the other ingredients in the investigational product.
24. Are unable or unwilling to withhold the use of eyelid scrubs or use of mechanical therapy during the study.
25. Have been diagnosed with glaucoma or are currently using any glaucoma medication.
26. Have a history of herpetic keratitis.
27. Have a concomitant ocular pathology other than condition under study assessed as potentially confounding by the investigator.
28. Have a serious systemic disease or uncontrolled medical condition that in the judgment of the investigator could confound study assessments or limit compliance.
29. Have been exposed to any investigational drug or investigational device within the preceding 30 days.
30. Are an employee of the site that is directly involved in the management, administration, or support of this study or be an immediate family member of the same.
31. Have trigger factors including conjunctivochalasis, allergic conjunctivitis, contact lens intolerance, trichiasis, epithelial basement membrane dystrophy, infectious keratitis or conjunctivitis.
32. Have a documented history of ocular allergies, which, in the judgment of the investigator, are likely to have an acute increase in severity due to the expected timing of the exposure to the allergen to which the subject is sensitive. Subjects sensitive to seasonal allergens that are not expected to be present during the study are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Vascular Engorgement in 1% HY02 Ointment compared to vehicle at week 12 | 12 Weeks
  Changes in Vascular Engorgement at the study eyelid margin are graded on a 5-point scale (0-4) with 0 representing minimal vascular engorgement and 4 representing maximal vascular engorgement. A lower score represents a better outcome for the subject.
Change from baseline in Eye Discomfort Visual Analogue Score (VAS) at week 12 in the 1% HY02 Ointment arm compared to vehicle | 12 Weeks
  Eye discomfort will be evaluated on a subject reported visual analog scale. The scores range from 0 (no discomfort) to 100 (maximal discomfort). Lower score indicate a better outcome for the subject.
Change from baseline in Vascular Engorgement in 0.3% HY02 Ointment compared to vehicle at week 12 | 12 Weeks
  Changes in Vascular Engorgement at the study eyelid margin are graded on a 5-point scale (0-4) with 0 representing minimal vascular engorgement and 4 representing maximal vascular engorgement. A lower score represents a better outcome for the subject.
Change from baseline in Eye Discomfort Visual Analogue Score (VAS) at week 12 in the 0.3% HY02 Ointment arm compared to vehicle | 12 Weeks
  Eye discomfort will be evaluated on a subject reported visual analog scale. The scores range from 0 (no discomfort) to 100 (maximal discomfort). Lower score indicate a better outcome for the subject.

CONTACTS AND LOCATIONS:
Overall Officials: George Magrath, MD, Study Director — Hovione Scientia Limited
Locations (20):
- United States (20):
  - Clinical site - 4, Azusa, California
  - Clinical site - 16, Huntington Beach, California
  - Clinical site - 12, Inglewood, California
  - Clinical site - 13, Mission Hills, California
  - Clinical site 10, Rancho Cordova, California
  - Clinical site - 15, Jacksonville, Florida
  - Clinical Site - 18, Largo, Florida
  - Clinical site - 6, Indianapolis, Indiana
  - Clinical site - 20, New Albany, Indiana
  - Clinical site - 19, Kansas City, Missouri
  - Clinical site - 3, St Louis, Missouri
  - Clinical site - 9, St Louis, Missouri
  - Clinical site - 7, Las Vegas, Nevada
  - Clinical site - 5, Asheville, North Carolina
  - Clinical site - 11, Mason, Ohio
  - Clinical site - 2, Memphis, Tennessee
  - Clinical site - 14, Cedar Park, Texas
  - Clinical Site - 1, El Paso, Texas
  - Clinical site - 8, League City, Texas
  - Clinical site - 17, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No